CLINICAL TRIAL: NCT02967484
Title: Acupuncture Lowering Blood Pressure for Secondary Prevention of Stroke: Study Protocol for a Multicenter, Pragmatic,Randomized Controlled, Assessor-blinded Clinical Trial
Brief Title: Acupuncture Lowering Blood Pressure for Secondary Prevention of Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Collaborators: State Administration of Traditional Chinese Medicine of the People's Republic of China (Other Government)
Responsible Party: Principal Investigator, Yuzheng Du, Director, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201507001-08
Record Dates: First submitted 2016-07-23; First posted 2016-11-18 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Cerebral Infarction
Keywords: Acupuncture; Hypertension; Second prevention of Stroke; Efficacy; RCT; Study protocol
MeSH Terms: conditions — Cerebral Infarction; Hypertension | interventions — Acupuncture Therapy; Dosage Forms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Participants will recieve the therapy as follows: "Huo Xue San Feng" acupuncture method+Routine care for ischemic stroke+One type of antihypertensive medication.
  Intervention:Acupuncture(choosing the bilatral acupoint: Renying(ST9),Hegu(L14), Taichong(LR3),Quchi(LI11),Zusanli(ST36))+Drugs(one type of antihypertensive medicine)
  Interventions: Device: acupuncture
- Control Group (No Intervention): Participants recieve the therapy as follows:Routine care for ischemic stroke +One type of antihypertensive medication.
  Intervention:Acupuncture(choosing the acupoint: Neiguan(PC6),Renzhong(10), Sanyinjiao(SP6),Jiquan(HT1),Chize(LU5),Weizhong(BL40).)+Drugs(one type of antihypertensive medicine)

INTERVENTIONS:
Device: acupuncture — 1. "Huo Xue San Feng" acupuncture method: Patients will recieve the acupuncture treatment,choose the bilateral point:Renying(ST9),Hegu(L14),Taichong(LR3),Quchi(LI11),Zusanli(ST36).
  2. Routine care for ischemic stroke :patients will recieve the acupuncture treatment,choose the point:Neiguan(PC6),Renzhong(10),Sanyinjiao(SP6),Jiquan(HT1),Chize(LU5),Weizhong(BL40).
  3. Drugs: Antihypertensive drugs.Patients will be treated 1 of 5 type of antihypertensive drugs,include ARB、ACEI、βreceptor blocker,CCB,Diuretic.
  The time of therapy will consist of 6 times per week in Continuous treatment phase(1st-6th week after enrollment) and 3 times per week(once every other day) in Consolidation treatment phase(7th-tewlve week after enrollment)
  Other Names: drug
  Arms: Treatment Group

SUMMARY:
This study evaluate the effects of acupuncture method on the recurrence of ischemic stroke patients.Half of participants will receive "Huo Xue San Feng" acupuncture combining 1 antihypertensive medication on the routine ischemic stroke treatments' basis. While the other half will receive 1 antihypertensive medication and basic treatments for ischemic stroke.

DETAILED DESCRIPTION:
Under recuiting 480 patients come from 5 hospitals in China.Eligible patients will be randomly assigned into 2 groups: treatment group and control group. The treatment group will receive "Huo Xue San Feng" acupuncture combining 1 antihypertensive medication on the routine ischemic stroke treatments' basis. The control group will receive 1 antihypertensive medication and basic treatments for ischemic stroke. "Huo Xue San Feng" acupuncture will be given six sessions weekly for the first 6 weeks and three times weekly for the next 6 weeks. A 9-month follow-up will thereafter be conducted. Antihypertensive medications will be adjusted based on BP levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the first time ischemic stroke
* Patients meet the TCM diagnosis standard of Stroke
* Patients meet the diagnosis standard of hypertension, taking only 1 type of antihypertensive drugs for at least 2 weeks before admission,corresponding to systolic pressure ranging from 140 to 160mmHg and Diastolic ranging from 90-100mmHg.
* The course of Ischemic stroke ranging from 2 weeks to 6 weeks .
* Men or Women Aged between 35 and 70 years old.
* Patients who are willing to participate in our clinical trial agree to sign the informed consent form.

Exclusion Criteria:

* Patients who have been diagnosed with secondary hypertension.
* Patients have taken beta blockers or diuretics or non dihydropyridine calcium channel blocker （NDHP-CCB）for a long time because of cardiovascular disease.
* Patients who taking 1 type of antihypertensive drugs,blood pressure under 140/90mmHg.
* Patients accompanied with other neurological disorders,such as epilepsy, peripheral nerve injury,
* Patients accompanied with severe medical condition such as severe hematopoietic system disease, coagulation dysfunction and malignant tumor.
* Patients accompanied with diabetic nephropathy,severe liver and renal insufficiency,severe cardiac or pulmonary dysfunction,severe arrhythmia.
* Patients who have occured skin infections near the acupoint location.
* Pregnant or breast-feeding women.
* Patients who currently participate in another clinical trial.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2016-11-20 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
The Effects of Acupuncture on Reccurence of Ischemic Stroke | 1 year after enrollment
  The effects of acupuncture on reccurence of ischemic stroke assessed by China's Guidelines of Diagnosis and Treatment of Acute Ischemic Stroke 2014 and China's Guidelines of Diagnosis and Treatment of Cerebral Hemorrhage 2014.

SECONDARY OUTCOMES:
24-hour ambulatory blood pressure | the first day、6 weeks、12 weeks after enrollment
Daily Blood Pressure by Electronic Sphygmomanometer | 1 year after enrollment
Antihypertensive Drug Stop/Resumption/Increasing Rate | 1 year after enrollment
Nitric Oxide(NO) | the first day、12 weeks,6 months after enrollment
Endothelin(ET) | the first day、12 weeks,6 months after enrollment
The Cardiac Color Doppler Ultrasonography | the first day、12 weeks after enrollment
Carotid Color Ultrasonography | the first day、12 weeks after enrollment
Brain Color Doppler Ultrasonography | the first day、12 weeks after enrollment
Lower Extremity Color Ultrasonography | the first day、12 weeks after enrollment
TCM syndrome score | the first day、6 weeks、12 weeks after enrollment
Short Form 36-item Health Survey (SF-36) | the first day、6 weeks、12 weeks after enrollment
National Institute of Health stroke scale (NIHSS)，as well as Barthel Index (BI) scale | the first day、12 weeks after enrollment
Essen stroke risk score (ESRS) | the first day、1 year after enrollment
All-caused Morality | 1 year after enrollment
Serum homocysteine（Hcy） | the first day、12 weeks,6 months after enrollment
Soluble CD40L（sCD40L） | the first day、12 weeks,6 months after enrollment
Copeptin | the first day、12 weeks,6 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Xuemin Shi, Study Director — The First Teaching Hospital of Tianjin University of TCM
Locations (5):
- China (5):
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing
  - MIANYANG Hospital of Traditional Chinese Medicine, Mianyang
  - LONGHUA Hospital Shanghai University of Traditional Chinese Medicine, Shanghai
  - Shenzhen Bao'an Traditional Chinese Medicine Hospital Group, Shenzhen
  - First Teaching Hospital of Tianjin University of TCM, Tianjin

REFERENCES:
- [Derived] Du YZ, Gao XX, Wang CT, Zheng HZ, Lei Y, Wu MH, Shi XM, Ban HP, Gu WL, Meng XG, Wei MT, Hu CX. Acupuncture lowering blood pressure for secondary prevention of stroke: a study protocol for a multicenter randomized controlled trial. Trials. 2017 Sep 15;18(1):428. doi: 10.1186/s13063-017-2171-5. PMID 28915826